CLINICAL TRIAL: NCT02487342
Title: Metabolic, Endocrine and Appetite-related Responses in Healthy, Adolescent Males After Acute and Daily Milk Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Dairy Council, United Kingdom (Other)
Responsible Party: Principal Investigator, Ben Green, Mr, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HLS-12-290413
Record Dates: First submitted 2015-06-18; First posted 2015-07-01 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Appetite Regulation
Keywords: Dairy; appetite; feeding behaviour
MeSH Terms: conditions — Feeding Behavior | interventions — Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- milk (Experimental): semi-skimmed milk (< 2% fat, Tesco, UK). All items were isovolumetric (217 mL) and isoenergetic (427 kJ).
  Interventions: Other: milk
- orange fruit-juice (Active Comparator): orange fruit-juice (Tesco, UK). All items were isovolumetric (217 mL) and isoenergetic (427 kJ).
  Interventions: Other: orange fruit-juice

INTERVENTIONS:
Other: milk — small serving (217 mL) of british semi-skimmed milk
  Arms: milk
Other: orange fruit-juice — small serving (217 mL) of orange juice
  Arms: orange fruit-juice

SUMMARY:
Comprising two experiments, the investigators assessed the metabolic, endocrine and appetite-related responses to acute (1-d, part 1) and daily mid-morning milk consumption (28-d, part 2) in adolescent males (15-18 y).

DETAILED DESCRIPTION:
The aims of the present study were twofold. Firstly, this study sought to examine the acute (1-d) effects of mid-morning milk consumption on subsequent metabolic, endocrine and appetite-related responses relative to an isoenergetic and isovolumetric serving of fruit-juice (part 1). Considering the putative mechanisms of milk consumption on appetite, feeding behavior and metabolism no studies are available that have explored the impact of daily milk or dairy food consumption on the above mentioned constructs in children and adolescents. This study therefore also aimed to compare the effect of daily (28-d) mid-morning milk or fruit-juice consumption on the above mentioned constructs (part 2).

Eleven adolescents participated in part 1 of this study and completed two trials (milk or fruit-juice mid-morning snack) in a randomized crossover design. For part 2, a parallel design with two intervention groups was employed. Participants were randomly allocated to groups, and received either a milk (n = 10) or an isocaloric and isovolumetric fruit-juice (n = 9) mid-morning snack for 28-d. On laboratory visits (for both part 1 and 2) participants remained at rest for 180 min. During this time, circulating concentrations of GLP-17-36, glucagon, insulin, leptin and blood glucose were determined. Measures of energy expenditure, substrate metabolism and subjective appetite were also collected. At 180 min, a homogenous ad libitum pasta meal was provided. For the remainder of the study day, subsequent energy intake was recorded utilizing a combined weighed self-reported food record and 24-h dietary recall technique.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Non diabetic
3. 15-18 yrs

Exclusion Criteria:

1. Are outside of the stipulated age range (15-18 years old)
2. A diabetic
3. Hold an aversion/dislike to milk, milk based products and the test meals provided.
4. Are known to be lactose intolerant
5. Currently taking any form of medication known to affect taste, smell and appetite
6. Female

Ages: 15 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Postprandial glucagon area under the curve | 180 min
  Fingertip-capillary measures of GLP-1 were collected at 30 min intervals throughout the 180 min protocol.

SECONDARY OUTCOMES:
Postprandial glucagonlike peptide-1 (GLP) area under the curve | 180 min
  Fingertip-capillary measures of glucagon were collected at 30 min intervals throughout the 180 min protocol.

OTHER OUTCOMES:
Postprandial insulin area under the curve | 180 min
  Fingertip-capillary measures of insulin were collected at 30 min intervals throughout the 180 min protocol.
Postprandial leptin area under the curve | 180 min
  Fingertip-capillary measures of insulin were collected at 30 min intervals throughout the 180 min protocol.
Postprandial blood glucose area under the curve | 180 min
  Fingertip-capillary measures of insulin were collected at 30 min intervals throughout the 180 min protocol.
Feeding behaviour | assessed at 180 min and following 24 h
  Energy intake was assessed at 180 min via an ad libitum pasta meal. Here subjects ate the pasta meal until they identified they were comfortably full. On completion of this, participants self-reported their energy intake for the remainder of the study day after leaving the laboratory.
Energy Expenditure | 180 min
  Measures of energy expenditure were calculated, through the use of Douglass Bags, for 300 seconds at 30 min intervals throughout the 180 min protocol.
Substrate oxidation | 180 min
  Measures of substrate oxidation were calculated, through the use of Douglass Bags, for 300 seconds at 30 min intervals throughout the 180 min protocol.
Subjective appetite | 180 min
  Subjective measures of appetite were collected at 30 min intervals throughout the 180 min protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin P Green, MSc, Principal Investigator — Northumbria University